CLINICAL TRIAL: NCT01344239
Title: Limb Remote Ischemic Preconditioning Reduces Heart and Lung Injury After Abdominal Aortic Aneurysm Repair:A Randomized Controlled Trial
Brief Title: Limb Remote Ischemic Preconditioning Reduces Heart and Lung Injury After Abdominal Aortic Aneurysm Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cai Li (Other)
Responsible Party: Sponsor-Investigator, Cai Li, Department of Anesthesiology,First Affiliated Hospital, Sun Yat-Sen University, Department of Anesthesiology,First Affiliated Hospital, Sun Yat-Sen University, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LRIP701126; CLi (Registry Identifier: CLi)
Record Dates: First submitted 2011-04-26; First posted 2011-04-29 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: aortic aneurysm; ischemia/reperfusion; preconditioning; pulmonary injury; intestinal injury
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm; Ischemia; Lung Injury

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Limb RIPC (Experimental): The limb RIPC protocol was applied after anesthetic induction and before the start of surgery. The limb RIPC was induced by placing a blood pressure cuff on the left upper arm of patient for three inflating-deflating cycles: 5 min inflating to 200 mmHg followed by a 5 min reperfusion with deflating the cuff.
  Interventions: Procedure: Limb remote ischemic preconditioning(LRIP)
- convention (No Intervention): Adult patients undergoing elective open abdominal aortic aneurysm repair received no treatment after induction of anaesthesia

INTERVENTIONS:
Procedure: Limb remote ischemic preconditioning(LRIP) — LRIP consisted of three cycles of left upper limb ischemia induced by inflating a blood pressure cuff on the left upper arm to 200mmHg, with an intervening 5 minutes of reperfusion, during which time the cuff was deflated.
  Other Names: LRIP
  Arms: Limb RIPC

SUMMARY:
To investigate whether limb remote ischemic preconditioning (LRIP) has protective effects against intestinal and pulmonary injury in patients undergoing open infrarenal abdominal aortic aneurysm (AAA) repair.

DETAILED DESCRIPTION:
Remote ischaemic preconditioning may confer the cytoprotection in critical organs. We hypothesized that limb remote ischemic preconditioning (RIPC) would reduce intestinal and pulmonary injury in patients undergoing open infrarenal abdominal aortic aneurysm (AAA) repair.The primary outcomes included the biomarkers reflecting intestinal injury (serum intestinal fatty acid binding protein, endotoxin levels and diamine oxidase activity) and the variables reflecting pulmonary injury (arterial-alveolar oxygen tension ratio, alveolar-arterial oxygen tension difference and respiratory index). In addition, the severity of intestinal and pulmonary injury was assessed with different scoring methods, respectively. Markers of oxidative stress and systemic inflammation were measured as well.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of abdominal aortic aneurysm
* Must be received open abdominal aortic aneurysm repair

Exclusion Criteria:

* age >80 years old
* Acute coronary syndrome or myocardial infraction within
* 3 months
* Chronic obstructive pulmonary emphysema
* angina pain within 48 hours of repair procedure
* ejection fraction less than 40%
* poor pulmonary function (PaO2 <60mmHg)
* history of inflammatory bowel disease
* history of diarrhea (≥2 liquid stools per day for ≥2 days) within 1 week of surgery
* intestinal chronic inflammatory disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-01; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Limb remote ischemic preconditioning has effective protection of lung injury in patients undergoing elective open abdominal aortic aneurysm repair | June,2011
  Compared with the control group, patients in the LRIP group had significantly higher Cs and Cd , along with lower PA-aDO2 and RI at various phase (P<0.05). Serum concentration of IL-6,IL-8, TNF-ɑ and MDA in LRIP group were decreased significantly at postoperative time points compared with those in control group (P<0.05), but SOD was increased significantly at the same time (P<0.05). Patient's ventilator support time and duration of ICU stay in LRIP group were shorter than that in control group (P<0.05)

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Xuan Liu, Ph.D, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University

REFERENCES:
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250